CLINICAL TRIAL: NCT05150574
Title: Pilot Testing a Health Coaching and Heart Rate Variability Biofeedback Program to Improve Stress and Well-being
Brief Title: HRV and Coaching Preparation Phase Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brock University (Other)
Collaborators: Mitacs (Industry)
Responsible Party: Principal Investigator, Sean Locke, Principal Investigator, Brock University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 20-367
Record Dates: First submitted 2021-11-15; First posted 2021-12-09 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Health Behavior; Work Related Stress; Job Stress; Anxiety Depression
Keywords: heart rate variability; health behaviour; anxiety; depression; job stress; well-being; health coaching
MeSH Terms: conditions — Health Behavior; Occupational Stress; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Condition 1 (Experimental): Core Health platform only
  Interventions: Behavioral: Core Health Program
- Condition 2 (Experimental): Core Health platform plus Practice with feedback coaching
  Interventions: Behavioral: Core Health Program; Behavioral: Practice with feedback coaching
- Condition 3 (Experimental): Core Health platform plus behavioural initiation coaching
  Interventions: Behavioral: Core Health Program; Behavioral: Behavioural initiation coaching
- Condition 4 (Experimental): Core Health platform plus Practice with feedback coaching and behavioural initiation coaching
  Interventions: Behavioral: Core Health Program; Behavioral: Behavioural initiation coaching; Behavioral: Practice with feedback coaching
- Condition 5 (Experimental): Core Health platform plus Momentary HRV feedback
  Interventions: Behavioral: Core Health Program; Behavioral: Momentary HRV feedback
- Condition 6 (Experimental): Core Health platform plus Momentary HRV feedback and Practice with feedback coaching
  Interventions: Behavioral: Core Health Program; Behavioral: Momentary HRV feedback; Behavioral: Practice with feedback coaching
- Condition 7 (Experimental): Core Health platform plus Momentary HRV feedback and behavioural initiation coaching
  Interventions: Behavioral: Core Health Program; Behavioral: Momentary HRV feedback; Behavioral: Behavioural initiation coaching
- Condition 8 (Experimental): Core Health platform plus Momentary HRV feedback, behavioural initiation coaching, and Practice with feedback coaching
  Interventions: Behavioral: Core Health Program; Behavioral: Momentary HRV feedback; Behavioral: Behavioural initiation coaching; Behavioral: Practice with feedback coaching
- Condition 9 (Experimental): Core Health platform plus Daily resting HRV
  Interventions: Behavioral: Core Health Program; Behavioral: Daily resting HRV
- Condition 10 (Experimental): Core Health platform plus Daily resting HRV feedback and Practice with feedback coaching
  Interventions: Behavioral: Core Health Program; Behavioral: Daily resting HRV; Behavioral: Practice with feedback coaching
- Condition 11 (Experimental): Core Health platform plus Daily resting HRV feedback and Behavioural initiation coaching
  Interventions: Behavioral: Core Health Program; Behavioral: Daily resting HRV; Behavioral: Behavioural initiation coaching
- Condition 12 (Experimental): Core Health platform plus Daily resting HRV feedback, Behavioural initiation coaching, and Practice with feedback coaching
  Interventions: Behavioral: Core Health Program; Behavioral: Daily resting HRV; Behavioral: Behavioural initiation coaching; Behavioral: Practice with feedback coaching
- Condition 13 (Experimental): Core Health platform plus Daily resting HRV feedback and Momentary HRV feedback
  Interventions: Behavioral: Core Health Program; Behavioral: Daily resting HRV; Behavioral: Momentary HRV feedback
- Condition 14 (Experimental): Core Health platform plus Daily resting HRV feedback, Momentary HRV feedback, and Practice with feedback coaching
  Interventions: Behavioral: Core Health Program; Behavioral: Daily resting HRV; Behavioral: Momentary HRV feedback; Behavioral: Practice with feedback coaching
- Condition 15 (Experimental): Core Health platform plus Daily resting HRV feedback, Momentary HRV feedback, and Behavioural initiation coaching
  Interventions: Behavioral: Core Health Program; Behavioral: Daily resting HRV; Behavioral: Momentary HRV feedback; Behavioral: Behavioural initiation coaching
- Condition 16 (Experimental): Core Health platform plus Daily resting HRV feedback, Momentary HRV feedback, Behavioural initiation coaching, and Practice with feedback coaching
  Interventions: Behavioral: Core Health Program; Behavioral: Daily resting HRV; Behavioral: Momentary HRV feedback; Behavioral: Behavioural initiation coaching; Behavioral: Practice with feedback coaching

INTERVENTIONS:
Behavioral: Core Health Program — 8-week structured stress management and health behaviour change program
Behavioral: Daily resting HRV — Take regular HRV readings in the morning
  Arms: Condition 10; Condition 11; Condition 12; Condition 13; Condition 14; Condition 15; Condition 16; Condition 9
Behavioral: Momentary HRV feedback — Take regular HRV readings throughout the day when stressed and perform mindfulness activity
  Arms: Condition 13; Condition 14; Condition 15; Condition 16; Condition 5; Condition 6; Condition 7; Condition 8
Behavioral: Behavioural initiation coaching — 15-minute health coaching session in first week of program to help participant set goals and create an action plan
  Arms: Condition 11; Condition 12; Condition 15; Condition 16; Condition 3; Condition 4; Condition 7; Condition 8
Behavioral: Practice with feedback coaching — 15-minute health coaching session in week 2 or 4 of program to help participant review goals and modify action plans if needed
  Arms: Condition 10; Condition 12; Condition 14; Condition 16; Condition 2; Condition 4; Condition 6; Condition 8

SUMMARY:
This pilot study will evaluate possible intervention components to be included in a future stress management and health behaviour change trial and to pilot test their feasibility and acceptability in a small sample.

DETAILED DESCRIPTION:
Work is one of the greatest contributors to chronic stress. Chronic stress is a critical risk factor leading to several negative work- and health-related outcomes. Developing scalable stress-management interventions will improve workers' health and wellness. The purpose of this project is to develop an optimized a stress reduction behavioural coaching and biofeedback intervention to supplement an existing mHealth platform (consisting of behavioural web-based modules). By testing coaching and biofeedback, this project can determine what level of interaction with a trained coach is necessary to optimally reduce workers' stress, and improve their health and well-being. To achieve this purpose, the multiphase optimization strategy (MOST) will be employed to develop, optimize, and evaluate the efficacy of this intervention. The three-phases include: preparation (selecting which intervention components are feasible to examine), optimization (determining the optimized package of components), and evaluation (evaluating the efficacy of the optimized package through a randomized control trial). This trial will cover the first phase of the MOST protocol. This pilot study will evaluate possible intervention components to be included in a future stress management and health behaviour change trial and to pilot test their feasibility and acceptability in a small sample.

Preparation phase objectives:

1.1 Determine which candidate components will be tested in a later optimization phase and at what dose they will be tested 1.2 Examine the feasibility of delivering the different components 1.3 Examine the acceptability of delivering the different components 1.4 Evaluate whether the outcomes can be feasibly measured

Design overview: A 2^4 (2x2x2x2) factorial experiment will run in the next phase of this project to test all combinations of four candidate components "turned on and off" with 16 different conditions. In the present study, we will ask 16 participants to each participate in and evaluate one of the sixteen conditions. The four candidate components being tested are: Daily resting HRV biofeedback, Momentary HRV biofeedback, Behavioural initiation coaching, and Practice with feedback coaching. Additionally, all participants will be asked to use complete the 8-week health behaviour change and stress management program on the Core health mHealth platform. Participants will be randomized to completing one of the sixteen conditions while completing the eight-week CoreHealth program.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Able to read and comprehend English
* Have smart phone (Android or iPhone 8 or higher)
* Self-report BMI under 40
* report at least Moderate daily stress

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Feasibility and acceptability of intervention components | Assessment taken immediately after the intervention
  Acceptability and Feasibility of Intervention Measure (Scale range 1[completely disagree] to 5 [completely agree] with higher scores being better; Weiner et al., 2017)
Participant perceptions of intervention components | Assessment taken immediately after the intervention
  Semi-structured interview questions to evaluate experiences, likes, dislikes, potential changes, and perceived feasibility
Health coach perceptions of intervention delivery | Assessment taken immediately after the intervention
  Semi-structured interview questions to evaluate experiences, likes, dislikes, potential changes, and perceived feasibility

SECONDARY OUTCOMES:
Heart rate variability | Assessment taken immediately before and after the intervention
  7-day device-measured HRV
Completion of survey measures | Assessment taken immediately before and after the intervention
  % of questionnaire measures answered and % missing data
User engagement | continuously collected during 8-week intervention
  number of times participants access the Core Health platform

CONTACTS AND LOCATIONS:
Overall Officials: Sean Locke, PhD, Principal Investigator — Brock University
Locations (1):
- Brock University, St. Catharines, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No